CLINICAL TRIAL: NCT05489770
Title: A Randomised, Single Blinded Study Investigating the Role of ' Black Elderberry (Sambucus Nigra) (Sambucol®) in the Treatment, Progression and Reduction of Symptoms in Participants With Coronavirus 19
Brief Title: BERRY- a Study of Sambucol ® in the Treatment, and Reduction of Symptoms in Participants With Coronavirus 19
Acronym: BERRY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: East Kent Hospitals University NHS Foundation Trust (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2020/COVID19/11
Record Dates: First submitted 2022-07-27; First posted 2022-08-05 (Actual); Results first posted 2024-12-06 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-10

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — Fluid Therapy

STUDY DESIGN:
Intervention Model Description: This study is a superiority test of Sambucol to placebo in the treatment of COVID 19 positive patients, with a parallel design.
  Single Centre, placebo controlled, single blinded, two arm, randomised controlled trial.
Who Masked: Participant, Outcomes Assessor
Masking Description: The placebo has comparable appearance and taste to Sambucol® Black Elderberry Original Liquid.
  Trial participants, trial statistician and outcome assessors will be blinded to which arm the participant has been randomised. Investigators, the research delivery team, clinical trial pharmacist and study staff not involved in assessing outcomes will not be blinded.
  All research delivery team members will be aware that they are not to divulge the randomised arm to participants at any time point.
  Participants will remain blind to their allocated trial arm for the duration of the trial.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sambucol® Black Elderberry Original (Sambucus nigra) Liquid (Active Comparator): Constituents: 29.4 % (w/w) Black Elderberry (Sambucus nigra) fruit juice, 70% (w/w) of glucose syrup.
  The main ingredient is black elderberry juice and it meets the requirements of the European Parliaments Directive (2012/12/EU) relating to fruit juices. The product also contains two food additives: citric acid (E330) as acidity regulator and potassium sorbate (E202) as preservative. Primary packaging: Plastic Polyethylene terephthalate (PET) amber bottles 120ml. Caps are white tamper-proof caps with security seal. Secondary Packaging: None. Outer Carton: Cardboard 376mm x 191mm x 116mm. 32 bottles per case.
  Interventions: Dietary Supplement: Sambucol® Black Elderberry Original (Sambucus nigra) Liquid
- Placebo for Sambucol® Black Elderberry Original (Sambucus nigra) Liquid (Placebo Comparator): Constituents: 70% (w/w) of glucose syrup, Flavouring agent: Elderberry Blossom. Colourants:
  Carmoisine (311804) (E-122) and Brilliant Black (419358) E-151. The product also contains two food additives: citric acid (E330) as acidity regulator and potassium sorbate (E202) as preservative. Primary packaging: Plastic PET amber bottles 120ml. Caps are white tamper-proof caps with security seal. Secondary Packaging: None. Outer Carton: Cardboard 376mm x 191mm x 116mm. 32 bottles per case.
  Interventions: Dietary Supplement: Placebo for Sambucol® Black Elderberry Original (Sambucus nigra)

INTERVENTIONS:
Dietary Supplement: Sambucol® Black Elderberry Original (Sambucus nigra) Liquid — Sambucol® Black Elderberry Original (Sambucus nigra) Liquid has been used as a supplement since 1991 with no reports of adverse effects received by the Manufacturer.
  Arms: Sambucol® Black Elderberry Original (Sambucus nigra) Liquid
Dietary Supplement: Placebo for Sambucol® Black Elderberry Original (Sambucus nigra) — Placebo for Sambucol® Black Elderberry Original (Sambucus nigra) Liquid Constituents: 70% (w/w) of glucose syrup, Flavouring agent: Elderberry Blossom
  Arms: Placebo for Sambucol® Black Elderberry Original (Sambucus nigra) Liquid

SUMMARY:
Severe acute respiratory syndrome (SARS) coronavirus 2 (CoV 2) (COVID19) is a readily transmissible virus that has a wide ranging incubation period of 2-14 days. The symptoms include fever, cough and loss of taste and smell. Symptoms range from mild to severe. Pre-existing potential drug therapies are under investigation, but so far few have demonstrated any benefit and only in patients with severe symptoms. There is a scarcity of other pre-existing drug treatments that change the outcomes/symptoms in non-hospitalised patients with COVID-19.

Prophylaxis and prevention is currently dependent on social distancing and isolating with vaccines remaining in development, potentially not for mass use in the near future.

Sambucus extract has well documented anti-viral properties both in vitro and in clinical trials of influenza, it has a low side effect profile so may be effective in reducing duration of symptoms and progression to more severe disease in patients with mild/ moderate COVID19. Black Elderberry Original Liquid (Sambucus nigra) (Sambucol®) is sold as a food supplement in heath food shops and supermarkets, does not require a prescription and has no known side effects, meaning it would be a well-tolerated treatment in early disease in comparison with other potential medications.

The study will be conducted at East Kent Hospitals. Potential participants with mild or moderate confirmed COVID19 infection will be identified from the drive-through hospital test centre and accident and emergency.

Following an eligibility check and consenting they would be randomised to placebo or Sambucol® Black Elderberry (Sambucus nigra) 15ml four times daily for 14 days which they will take at home. Telephone consultations with the research team and patient daily diaries will used to document symptoms on days 1,3,7,10,14 and a follow up on day 28. Time to clinical improvement will be compared between the 2 groups.

DETAILED DESCRIPTION:
The outbreak of the new coronavirus SARS-CoV-2 (COVID-19) in China has rapidly progressed to pandemic status of global importance. The current lack of a proven anti-viral that is effective has meant the current management of severe respiratory coronaviruses remains supportive. The success achieved in treating bacterial infections is not paralleled in antivirals. The relative paucity lies in a lack of drugs that stop replication within a living cell, and that the peak rate of growth may occur prior to symptoms.

A randomised controlled trial of lopinavir/ritonavir (an antiviral treatment commonly used to treat HIV) compared to standard of care in patients with severe COVID-19 demonstrated no clinical benefit and in 13.8% treatment had to be stopped early due to adverse events . Prophylactic use of hydroxychloroquine continues worldwide both within and outside of clinical trials but concern remains with prescribing an unproven drug with well-known adverse neurological and cardiac effects .'RECOVERY' is a large United Kingdom (UK) randomised controlled trial established to test a range of potential treatments for COVID-19 in hospitalised patients, including lopinavir/ritonavir and hydroxychloroquine. Over 12,000 patients have been enrolled from 176 National Health Service (NHS) hospitals. It showed no benefit of hydroxychloroquine nor lopinavir/ritonavir in this population, and by contrast, that low-dose dexamethasone reduces the risk of death by about one-third among patients receiving ventilation and by one-fifth in those requiring oxygen alone. However, no benefit was demonstrated amongst those not requiring respiratory support. Pharmacognosy is the study of medicines derived from natural sources. Plant extracts have been widely used to treat a number of medical conditions, with some of the best-known examples including, quinine isolated from Cinchona pubescens (cinchona tree) used to treat malaria, Papaver somniferum to make morphine and Digitalis purpurea for treating atrial fibrillation. A number of plant constituents have demonstrated anti-viral activity. Hippocrates, 'Father of Medicine' referred to Elderberry as 'natures medicine chest'.

In vitro Sambucus Formosana Nakai extract showed potent antiviral activity against human coronavirus Netherlands 63 ( NL63) in terms of decreased cytopathic effect and sub-G1 arrest in coronavirus infected cells. It produces a significant reduction in viral yield, plaque formation and virus attachment. The authors conclude that like Sambucus nigra L., Sambucus FormosanaNakai might possess antiviral features against the broad spectrum of human respiratory coronaviruses . This supports the previously published data of Sambucus spp., and Sambucus nigra L. providing the antiviral properties against influenza A and B viruses and herpes simplex type 1 . In 1995 it was demonstrated a significant improvement in symptoms in 93.3% of patients treated with standardised elderberry extract within 2 days compared to within 6 days in the control arm (p<0.001).

Complete cure occurred in 90% of those receiving the extract in 2 to 3 days . Subsequent randomised double -blind studies demonstrated no adverse events and significant improvement in clinical symptoms and higher antibody titres in those receiving Sambuci fructus .Chen at al 2014 demonstrated with in vitro testing of coronavirus Infectious Bronchitis Virus (IBV) with Sambucus.nigra a reduction in virus titres by four orders of magnitude, compromised envelopes and membrane vesicles. This virion disruption likely renders it non-infectious . Of further interest was that complete inhibition occurred when pre-treatment of virus in combination with post- infection treatment.

SARS-CoV-2 (COVID-19) is a readily transmissible virus that has a wide-ranging incubation period of 2-14 days (US Centers for Disease Control and Prevention). The symptoms are often non-specific and include fever, cough, fatigue, diarrhoea and loss of sense of taste and smell. Clinical features range from mild to severe. Varying transmission patterns and mild symptoms are of concern as they facilitate rapid spread. Pre-existing potential drug therapies are under investigation, and only started once the patient has symptoms, but do have well established side effect profiles. Prophylaxis and prevention are currently dependent on social distancing and isolating with vaccines remaining in development, potentially not for mass use in the near future.

Sambucus extract has well documented anti-viral properties and no known drug interactions were identified in the literature. Hence, Sambucus maybe well suited for limited prophylaxis or treatment of mild/ moderate COVID-19. There is clear in Vitro evidence of activity against coronavirus and in human trials of influenza. The aim of this study is to see if Sambucol® Black Elderberry Original Liquid (Sambucus nigra) at a dose of 15ml, 4 times a day, reduces the duration or severity of symptoms of COVID-19. Symptomatic patients presenting to drive through testing (i.e. non-hospitalised) who test positive and who consent will be randomised to placebo or Sambucol® and blinded to treatment allocation. Study staff/investigators responsible for assessing outcomes and data analysis will also be blinded to treatment allocation. Data will be collected to determine resolution of symptoms and the two groups compared.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic Severe acute respiratory syndrome coronavirus 2 (SARS-CoV2) infection
* Positive SARS-CoV2 swab test result within the last 5 days
* Capacity to provide written or electronic informed consent
* Able to complete follow up visits required via phone/email
* Able to provide a positive swab result

Exclusion Criteria:

Known allergy to Sambucus (Elderberries) or food colourants

* Pregnant or breast feeding
* Poorly controlled diabetes
* Treatment with any immunosuppressive medicines including Prednisolone 10mg daily or equivalent. Oral anti-inflammatory medicines such as Ibuprofen are allowed.
* Participation in any COVID 19 research study involving prophylactic or therapeutic Investigational Medicinal Products (IMPs) in the last 30 days.
* Previous participation in this trial.
* Already taking Sambucol or any form of elderberry supplement

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 204 (Actual)
Dates: Start 2021-01-05 (Actual); Primary Completion 2022-05-16 (Actual); Study Completion 2022-05-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jessica Evans, Principal Investigator — EKHUFT
Locations (1):
- East Kent Hospitals University NHS Foundation trust, Canterbury, Kent, United Kingdom

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Sambucol® Black Elderberry Original (Sambucus Nigra) Liquid: Constituents: 29.4 % (w/w) Black Elderberry (Sambucus nigra) fruit juice, 70% (w/w) of glucose syrup.
  The main ingredient is black elderberry juice and it meets the requirements of the European Parliaments Directive (2012/12/EU) relating to fruit juices. The product also contains two food additives: citric acid (E330) as acidity regulator and potassium sorbate (E202) as preservative. Primary packaging: Plastic Polyethylene terephthalate (PET) amber bottles 120ml. Caps are white tamper-proof caps with security seal. Secondary Packaging: None. Outer Carton: Cardboard 376mm x 191mm x 116mm. 32 bottles per case.
  Sambucol® Black Elderberry Original (Sambucus nigra) Liquid: Sambucol® Black Elderberry Original (Sambucus nigra) Liquid has been used as a supplement since 1991 with no reports of adverse effects received by the Manufacturer.
- Placebo for Sambucol® Black Elderberry Original (Sambucus Nigra) Liquid: Constituents: 70% (w/w) of glucose syrup, Flavouring agent: Elderberry Blossom. Colourants:
  Carmoisine (311804) (E-122) and Brilliant Black (419358) E-151. The product also contains two food additives: citric acid (E330) as acidity regulator and potassium sorbate (E202) as preservative. Primary packaging: Plastic PET amber bottles 120ml. Caps are white tamper-proof caps with security seal. Secondary Packaging: None. Outer Carton: Cardboard 376mm x 191mm x 116mm. 32 bottles per case.
  Placebo for Sambucol® Black Elderberry Original (Sambucus nigra): Placebo for Sambucol® Black Elderberry Original (Sambucus nigra) Liquid Constituents: 70% (w/w) of glucose syrup, Flavouring agent: Elderberry Blossom
Period: Overall Study
Arm/Group | Sambucol® Black Elderberry Original (Sambucus Nigra) Liquid | Placebo for Sambucol® Black Elderberry Original (Sambucus Nigra) Liquid
Started | 102 | 102
Completed | 93 | 90
Not Completed | 9 | 12

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sambucol® Black Elderberry Original (Sambucus Nigra) Liquid | Placebo for Sambucol® Black Elderberry Original (Sambucus Nigra) Liquid | Total
Number analyzed (Participants) | 102 | 102 | 204
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 100 | 101 | 201
  >=65 years | 2 | 1 | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 64 | 73 | 137
  Male | 38 | 29 | 67
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  white | 96 | 94 | 190
  Asian | 5 | 5 | 10
  Mixed/Other | 1 | 3 | 4
Region of Enrollment [Number; unit: participants]
  United Kingdom | 102 | 102 | 204
Wellness score at day 0 [Mean (Standard Deviation); unit: units on a scale (0-100)] — The scale used went from 0-100. where 0- worst health, 100 best health. Patients described what value they felt their pain was at each time point
  units on a scale (0-100) | 60.9 (20.5) | 60.7 (17.9) | 60.8 (19)

OUTCOME MEASURES:

1. Primary Outcome: Sambucol Reduces the Severity of Symptoms by at Least 30% by Day 10 in People Who Are Symptomatic With the SARS-CoV-2 (COVID-19) Virus, Compared to Placebo.
Description: To determine whether Sambucol reduces the severity of symptoms by 30% by day 10 in people who are symptomatic with the COVID-19 virus, as determined by Visual Analogue Scale score. where 0 was worst health and 100 best health
Time Frame: 10 days
Population: VAS score where 100 is best health and 0 is worst. AT this time point there were 90 participants who replied in the "test" group and 93 in the placebo
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Sambucol® Black Elderberry Original (Sambucus Nigra) Liquid | Placebo for Sambucol® Black Elderberry Original (Sambucus Nigra) Liquid
Number analyzed (Participants) | 90 | 93
score on a scale | 84.3 (13.8) | 86.5 (9.9)

2. Secondary Outcome: To Determine Whether Sambucol Reduces Hospital Admissions by Day 28.
Description: To determine whether Sambucol reduces number of hospital admissions by day 28.
Time Frame: 28 days
Population: No hospital admissions in either group
Measure: Count of Participants; unit: Participants
Arm/Group | Sambucol® Black Elderberry Original (Sambucus Nigra) Liquid | Placebo for Sambucol® Black Elderberry Original (Sambucus Nigra) Liquid
Number analyzed (Participants) | 84 | 87
Participants | 0 | 0

3. Secondary Outcome: To Determine if Sambucol Reduces the Severity of Symptoms at Day 3, 7, 14 and 28 Days
Description: To determine if Sambucol reduces the severity of symptoms at day 3, 7, 14 and 28 days as determined by a Visual Analogue Scale _(VAS) where 0 was worst health and 100 best health
Time Frame: 28 days
Population: The number analysed at each time point varies as not all participants replied at each time point
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Sambucol® Black Elderberry Original (Sambucus Nigra) Liquid | Placebo for Sambucol® Black Elderberry Original (Sambucus Nigra) Liquid
Number analyzed (Participants) | 102 | 102
score on a scale
  Day 3: number analyzed (Participants) | 101 | 96
  Day 3 | 68.6 (19.5) | 68.6 (15.6)
  Day 7: number analyzed (Participants) | 96 | 96
  Day 7 | 78.9 (17) | 80.3 (12.7)
  DAy 14: number analyzed (Participants) | 90 | 92
  DAy 14 | 88.7 (13.9) | 91.1 (8.8)
  Day 28: number analyzed (Participants) | 84 | 87
  Day 28 | 93.5 (11.4) | 94.8 (7.1)

4. Other Pre Specified Outcome: Reduction in Hospital Admission as Per Participant Hospital Admission Rates
Description: Reduction in hospital admission as per participant hospital admission rates- for participants with mild or moderate COVID-19
Time Frame: 28 days
Population: How many participants were admitted to hospital
Measure: Count of Participants; unit: Participants
Arm/Group | Sambucol® Black Elderberry Original (Sambucus Nigra) Liquid | Placebo for Sambucol® Black Elderberry Original (Sambucus Nigra) Liquid
Number analyzed (Participants) | 84 | 87
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: Each participant was in the trial for 28 days , adverse event data will be collected over this period- 28 days
Arm/Group | Sambucol® Black Elderberry Original (Sambucus Nigra) Liquid | Placebo for Sambucol® Black Elderberry Original (Sambucus Nigra) Liquid
All-Cause Mortality (participants affected / at risk) | 0/102 | 0/102
Serious Adverse Events (participants affected / at risk) | 1/102 | 0/102
Other Adverse Events (participants affected / at risk) | 19/102 | 16/102
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sambucol® Black Elderberry Original (Sambucus Nigra) Liquid (N=102) | Placebo for Sambucol® Black Elderberry Original (Sambucus Nigra) Liquid (N=102)
Shortness of breath and chest pain (Respiratory, thoracic and mediastinal disorders) | 1 | NA
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Sambucol® Black Elderberry Original (Sambucus Nigra) Liquid (N=102) | Placebo for Sambucol® Black Elderberry Original (Sambucus Nigra) Liquid (N=102)
skin (Skin and subcutaneous tissue disorders) | 7 | 5
Gastro (Gastrointestinal disorders) | 5 | 4
general (General disorders) | 7 | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-07-22): https://cdn.clinicaltrials.gov/large-docs/70/NCT05489770/Prot_SAP_000.pdf